CLINICAL TRIAL: NCT03564002
Title: Metabolic Effects of Very Low Carbohydrate Ketogenic Diet in Subjects With Severe Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Maria Anastasia Ricci, Principal Investigator, University Of Perugia
Other Study IDs: 2017-12
Record Dates: First submitted 2018-05-26; First posted 2018-06-20 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Lysosomal Acid Lipase Deficiency; Obesity; Ketogenic Dieting; Ketosis
MeSH Terms: conditions — Wolman Disease; Obesity; Ketosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese subjects
- lean subjects

SUMMARY:
The very low carbohydrates diet (VLCKD) induces liver steatosis amelioration. Lysosomal acid lipase (LAL) deficiency plays a role in fats accumulation in liver. To date, no studies have assessed LAL activity in morbid obesity. The aim of our study is to evaluate VLCKD impact on metabolic/vascular parameters and LAL activity in obese patients.

A VLCKD is administered for 25 days to 52 morbid obese patients (BMI 44.7±8.3 kg/m², age 49±12.5 years); at baseline and after diet we evaluated: BMI, glyco-lipidic pattern, abdominal ultrasonography (liver steatosis and visceral fat area) and flow-mediated dilation (FMD). In a subgroup of 20 patients we also tested lysosomal acid lipase (LAL)-activity. A group of healthy normal weight subjects (age 43±13, BMI 22.8±2.6 kg/m²) was also included in the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 Kg/m2 or > 35 kg/m2 with comorbidities

Exclusion Criteria:

* Type-2 diabetes
* Kidney, heart or liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese patients referred to our Clinic in order to assess and treat obesity
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
lysosomal acid lipase activity | change from baseline after 25 days
  LAL-activity was dosed with dried blood spot (DBS) technique using the inhibitors Lalistat 2
endothelial function | change from baseline after 25 days
  flow mediated dilation at brachial artery by ultrasonography
visceral fat | change from baseline after 25 days
  ultrasonography
liver steatosis | change from baseline after 25 days
  ultrasonography
lipid assessment | change from baseline after 25 days
  total cholesterol, triglycerides, HDL, LDL
general adiposity assessment | change from baseline after 25 days
  bioimpedentiometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Perugia, Perugia, Italy